CLINICAL TRIAL: NCT02600494
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Multi-Center Study With an Open-Label Extension to Assess the Efficacy and Safety of ITI-007 Monotherapy in the Treatment of Patients With Major Depressive Episodes Associated With Bipolar I or Bipolar II Disorder (Bipolar Depression)
Brief Title: Clinical Trial Evaluating ITI-007 (Lumateperone) as a Monotherapy for the Treatment of Bipolar Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Intra-Cellular Therapies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ITI-007-401
Record Dates: First submitted 2015-11-05; First posted 2015-11-09 (Estimated); Results first posted 2025-11-03 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Bipolar Depression
MeSH Terms: conditions — Bipolar Disorder | interventions — lumateperone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 40 mg ITI-007 (Lumateperone) (Experimental): 40 mg ITI-007 (Lumateperone) administered orally as capsules once daily for 6 weeks
  Interventions: Drug: ITI-007 (Lumateperone)
- 60 mg ITI-007 (Lumateperone) (Experimental): 60 mg ITI-007 (Lumateperone) administered orally as capsules once daily for 6 weeks
  Interventions: Drug: ITI-007 (Lumateperone)
- Placebo (Placebo Comparator): Placebo administered orally as visually-matched capsules once daily for 6 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ITI-007 (Lumateperone)
  Arms: 40 mg ITI-007 (Lumateperone); 60 mg ITI-007 (Lumateperone)
Drug: Placebo
  Arms: Placebo

SUMMARY:
The study will evaluate the efficacy and safety of ITI-007 (Lumateperone) in patients diagnosed with Bipolar I or Bipolar II disorder having a major depressive episode. The study will be conducted in two parts, Part A and Part B. Part A is a randomized, double-blind, placebo-controlled study. In Part B, patients who safely complete participation in part A may be enrolled in an open-label extension.

ELIGIBILITY:
Major Inclusion Criteria:

* male or female subjects of any race, ages 18-75 inclusive, with a clinical diagnosis of Bipolar I or Bipolar II disorder
* experiencing a current major depressive episode

Major Exclusion Criteria:

* any subject unable to provide informed consent
* any female subject who is pregnant or breast-feeding
* any subject judged to be medically inappropriate for study participation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 554 (Actual)
Dates: Start 2015-12-15 (Actual); Primary Completion 2019-01-28 (Actual); Study Completion 2019-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Kozauer, MD, Study Director — Intra-Cellular Therapies, Inc. (ITI)
Locations (55):
- United States (55):
  - Clinical Site, Little Rock, Arkansas
  - Clinical Site, Rogers, Arkansas
  - Clinical Site, Cerritos, California
  - Clinical Site, Culver City, California
  - Clinical Site, Garden Grove, California
  - Clinical Site, Lemon Grove, California
  - Clinical Site, National City, California
  - Clinical Site, Oakland, California
  - Clinical Site, Oceanside, California
  - Clinical Site, Orange, California
  - Clinical Site, Pico Rivera, California
  - Clinical Site, Riverside, California
  - Clinical Site, San Diego, California
  - Clinical Site, San Marcos, California
  - Clinical Site, Santa Rosa, California
  - Clinical Site, Colorado Springs, Colorado
  - Clinical Site, Bradenton, Florida
  - Clinical Site, Fort Myers, Florida
  - Clinical Site, Jacksonville, Florida
  - Clinical Site, Lauderhill, Florida
  - Clinical Site, Miami, Florida
  - Clinical Site, North Miami, Florida
  - Clinical Site, Orlando, Florida
  - Clinical Site, Atlanta, Georgia
  - Clinical Site, Chicago, Illinois
  - Clinical Site, Hoffman Estates, Illinois
  - Clinical Site, Lake Charles, Louisiana
  - Clinical Site, Baltimore, Maryland
  - Clinical Site, Boston, Massachusetts
  - Clinical Site, O'Fallon, Missouri
  - Clinical Site, St Louis, Missouri
  - Clinical Site, Las Vegas, Nevada
  - Clinical Site, Berlin, New Jersey
  - Clinical Site, Cherry Hill, New Jersey
  - Clinical Site, Marlton, New Jersey
  - Clinical Site, Toms River, New Jersey
  - Clinical Site, Brooklyn, New York
  - Clinical Site, Cedarhurst, New York
  - Clinical Site, New York, New York
  - Clinical Site, Rochester, New York
  - Clinical Site, Staten Island, New York
  - Clinical Site, Cincinnati, Ohio
  - Clinical Site, Cleveland, Ohio
  - Clinical Site, Dayton, Ohio
  - Clinical Site, Garfield Heights, Ohio
  - Clinical Site, Oklahoma City, Oklahoma
  - Clinical Site, Allentown, Pennsylvania
  - Clinical Site, Norristown, Pennsylvania
  - Clinical Site, Philadelphia, Pennsylvania
  - Clinical Site, Memphis, Tennessee
  - Clinical Site, Austin, Texas
  - Clinical Site, Dallas, Texas
  - Clinical Site, Houston, Texas
  - Clinical Site, Petersburg, Virginia
  - Clinical Site, Everett, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Part A includes all patients who signed the informed consent and were randomized in to the 6 week double-blind treatment period. 554 patients were randomized; 549 patients received study drug and are included in the safety population.
  Part B includes all patients who signed the informed consent and received open-label study drug for up to 6 months.
Groups:
- Lumateperone 28 mg (ITI-007 40 mg Tosylate): Lumateperone 28 mg (ITI-007 40 mg tosylate) administered orally as capsules once daily for 6 weeks
  ITI-007 (Lumateperone)
- Lumateperone 42 mg (ITI-007 60 mg Tosylate): Lumateperone 42 mg (ITI-007 60 mg tosylate) administered orally as capsules once daily for 6 weeks
  Lumateperone (ITI-007)
- Placebo: Placebo administered orally as visually-matched capsules once daily for 6 weeks
  Placebo
Period: Part A (6 Week Double-Blind Treatment)
Arm/Group | Lumateperone 28 mg (ITI-007 40 mg Tosylate) | Lumateperone 42 mg (ITI-007 60 mg Tosylate) | Placebo
Started | 183 | 185 | 186
Number of Patients Randomized and Took at Least 1 Dose of Study Drug | 180 | 184 | 185
Completed | 126 | 113 | 138
Not Completed | 57 | 72 | 48
Not completed — Adverse Event | 13 | 15 | 4
Not completed — Lack of Efficacy | 2 | 4 | 2
Not completed — Protocol Violation | 13 | 10 | 14
Not completed — Physician Decision | 2 | 3 | 4
Not completed — Withdrawal by Subject | 15 | 11 | 14
Not completed — Lost to Follow-up | 12 | 28 | 10
Not completed — non-compliant with site request | 0 | 1 | 0
Period: Part B (6 Month Open-Label Treatment)
Arm/Group | Lumateperone 28 mg (ITI-007 40 mg Tosylate) | Lumateperone 42 mg (ITI-007 60 mg Tosylate) | Placebo
Started | 0 (This was an open label portion of the study where all pts received Lumateperone 42 mg/day; therefore, the Lumateperone 28 mg and Placebo arms are not applicable.) | 127 (For some patients Part B was not a direct rollover; therefore, the number of patients that completed Part A does not equal the number of patients enrolled in Part B.) | 0 (This was an open label portion of the study where all pts received Lumateperone 42 mg/day; therefore, the Lumateperone 28 mg and Placebo arms are not applicable.)
Completed | 0 | 74 | 0
Not Completed | 0 | 53 | 0
Not completed — Adverse Event | 0 | 12 | 0
Not completed — Lack of Efficacy | 0 | 4 | 0
Not completed — Protocol Violation | 0 | 8 | 0
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 17 | 0
Not completed — Lost to Follow-up | 0 | 11 | 0

BASELINE CHARACTERISTICS:
Population: All patients in Part A Safety Analysis set which contains all patients who received at least one dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Lumateperone 28 mg (ITI-007 40 mg Tosylate) | Lumateperone 42 mg (ITI-007 60 mg Tosylate) | Placebo | Total
Number analyzed (Participants) | 180 | 184 | 185 | 549
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.5 (12.12) | 42.7 (11.85) | 42.3 (13.13) | 41.9 (12.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109 | 111 | 114 | 334
  Male | 71 | 73 | 71 | 215
Race/Ethnicity, Customized [Number; unit: participants]
  White | 100 | 106 | 98 | 304
  Black or African American | 75 | 72 | 80 | 227
  Asian | 1 | 2 | 3 | 6
  American Indian or Alaska Native | 0 | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1 | 2
  Multiple | 4 | 1 | 1 | 6
  Not Reported | 0 | 0 | 1 | 1
Montgomery Asberg Depression Rating Scale (MADRS) [Mean (Standard Deviation); unit: units on a scale] | 35.8 (6.08) | 35.9 (5.79) | 34.7 (5.84) | 35.4 (5.92)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Day 43 in Montgomery-Åsberg Depression Rating Scale (MADRS) Total Score
Description: The Montgomery-Åsberg Depression Rating Scale (MADRS) is a clinician-rated 10 item scale to assess depressive symptoms. Each item is rated on a 7-point scale from 0-6. The total score ranges from 0 to 60 with a higher score indicating increased severity of depressive symptoms.
Time Frame: 6 weeks
Population: Intent-to-Treat (ITT) Set contains all randomized patients who received at least one dose of study medication and who had a valid baseline (pre-dose) measurement and at least one valid post-baseline measurement of MADRS total score.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Lumateperone 28 mg (ITI-007 40 mg Tosylate) | Lumateperone 42 mg (ITI-007 60 mg Tosylate) | Placebo
Number analyzed (Participants) | 172 | 166 | 177
score on a scale | -18.9 (1.11) | -20.7 (1.16) | -19.7 (1.11)
Statistical Analysis 1: Comparison: Lumateperone 28 mg (ITI-007 40 mg Tosylate) vs Placebo; Test type: Superiority; p = 0.514, Mixed Effects Model for Repeated Measure — p-value is Hochberg-adjusted; Least Squares Mean Difference = 0.9, 95% CI 2-sided [-1.83 to 3.53]
Statistical Analysis 2: Comparison: Lumateperone 42 mg (ITI-007 60 mg Tosylate); Test type: Superiority; p = 0.895, Mixed Effects Model for Repeated Measure — p-value is Hochberg adjusted; Least Squares Mean Difference = -1.0, 95% CI 2-sided [-3.73 to 1.79]

2. Secondary Outcome: Time to First Sustained Response in Reduction of MADRS Total Score
Time Frame: 6 weeks
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Lumateperone 28 mg (ITI-007 40 mg Tosylate) | Lumateperone 42 mg (ITI-007 60 mg Tosylate) | Placebo
Number analyzed (Participants) | 172 | 166 | 177
days | 43 [36 to NA] — Upper limit of the confidence interval could not be calculated due to insufficient number of events. | 38 [36 to NA] — Upper limit of the confidence interval could not be calculated due to insufficient number of events. | 37 [30 to NA] — Upper limit of the confidence interval could not be calculated due to insufficient number of events.
Statistical Analysis 1: Comparison: Lumateperone 28 mg (ITI-007 40 mg Tosylate) vs Placebo; Test type: Superiority; p = 0.993, Regression, Cox; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.712 to 1.400]
Statistical Analysis 2: Comparison: Lumateperone 42 mg (ITI-007 60 mg Tosylate) vs Placebo; Test type: Superiority; p = 0.665, Regression, Cox; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.657 to 1.307]

3. Other Pre Specified Outcome: Change From Baseline to Day 175 in Montgomery-Åsberg Depression Rating Scale (MADRS) Total Score
Description: The MADRS total score from baseline to Day 175 for patients that rolled over into the extension portion of the study (Part B)
Time Frame: Day 175
Population: Safety Analysis Set - all patients who received at least 1 dose of study medication in Part B
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Lumateperone 42 mg (ITI-007 60 mg Tosylate): Lumateperone 42 mg (ITI-007 60 mg tosylate) administered orally as capsules once daily for approximately 6 months
Arm/Group | Lumateperone 42 mg (ITI-007 60 mg Tosylate)
Number analyzed (Participants) | 127
units on a scale | -8.9 (10.76)

4. Other Pre Specified Outcome: Adverse Events
Description: Incidence of Treatment-Emergent Adverse Events from baseline to Day 175 for patients that rolled over into the extension portion of the study (Part B)
Time Frame: Day 175
Measure: Count of Participants; unit: Participants
Arm/Group | Lumateperone 42 mg (ITI-007 60 mg Tosylate)
Number analyzed (Participants) | 127
Participants
  Headache | 26
  Dry Mouth | 15
  Dizziness | 13
  Nausea | 13
  Somnolence | 11
  Anxiety | 10
  Irritability | 8

ADVERSE EVENTS:
Time Frame: From signing ICF until end of study procedures (~10 weeks), including 6 weeks of double-blind treatment
Groups:
- Part A Lumateperone 28 mg (ITI-007 40 mg Tosylate): Lumateperone 28 mg (ITI-007 40 mg tosylate) administered orally as capsules once daily for 6 weeks
  ITI-007 (Lumateperone)
- Part A Lumateperone 42 mg (ITI-007 60 mg Tosylate): Lumateperone 42 mg (ITI-007 60 mg tosylate) administered orally as capsules once daily for 6 weeks
  Lumateperone (ITI-007)
- Part A Placebo: Placebo administered orally as visually-matched capsules once daily for 6 weeks
  Placebo
- Part B Lumateperone 42 mg (ITI-007 60 mg Tosylate): Lumateperone 42 mg (ITI-007 60 mg tosylate) administered orally as capsules once daily for up to 6 months
  Lumateperone (ITI-007)
Arm/Group | Part A Lumateperone 28 mg (ITI-007 40 mg Tosylate) | Part A Lumateperone 42 mg (ITI-007 60 mg Tosylate) | Part A Placebo | Part B Lumateperone 42 mg (ITI-007 60 mg Tosylate)
All-Cause Mortality (participants affected / at risk) | 0/180 | 0/184 | 1/185 | 0/127
Serious Adverse Events (participants affected / at risk) | 5/180 | 0/184 | 1/185 | 4/127
Other Adverse Events (participants affected / at risk) | 72/180 | 67/184 | 31/185 | 55/127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A Lumateperone 28 mg (ITI-007 40 mg Tosylate) (N=180) | Part A Lumateperone 42 mg (ITI-007 60 mg Tosylate) (N=184) | Part A Placebo (N=185) | Part B Lumateperone 42 mg (ITI-007 60 mg Tosylate) (N=127)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Mania (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Panic Attack (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicidal Ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Agression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anemia postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Procedural hemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
colitis ulcerative (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A Lumateperone 28 mg (ITI-007 40 mg Tosylate) (N=180) | Part A Lumateperone 42 mg (ITI-007 60 mg Tosylate) (N=184) | Part A Placebo (N=185) | Part B Lumateperone 42 mg (ITI-007 60 mg Tosylate) (N=127)
Somnolence (Nervous system disorders) | 21 | 24 | 7 | 11
Headache (Nervous system disorders) | 35 | 20 | 10 | 26
Nausea (Gastrointestinal disorders) | 12 | 16 | 7 | 13
Dry Mouth (Gastrointestinal disorders) | 13 | 15 | 3 | 15
Dizziness (Nervous system disorders) | 10 | 15 | 4 | 13
Diarrhoea (Gastrointestinal disorders) | 9 | 10 | 5 | 4
Vomiting (Gastrointestinal disorders) | 5 | 10 | 0 | 6
Fatigue (General disorders) | 11 | 4 | 3 | 4
Anxiety (Psychiatric disorders) | 1 | 2 | 3 | 10
Irritability (Psychiatric disorders) | 3 | 3 | 1 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-03-09): https://cdn.clinicaltrials.gov/large-docs/94/NCT02600494/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-12): https://cdn.clinicaltrials.gov/large-docs/94/NCT02600494/SAP_001.pdf